CLINICAL TRIAL: NCT06561282
Title: The Predictive Role of Glucose/Potassium Ratio for Mortality in Patients With Major Burn Trauma
Brief Title: Predictive Role of Glucose/Potassium Ratio on Mortality in Major Burns.
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, Principal investigator, Konya Meram State Hospital
Other Study IDs: Konya Burn Center
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burns; Burn Injury; Inhalation Injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to investigate the role of the glucose-potassium ratio in predicting mortality in patients with major burn trauma.

The main question it aims to answer is: Can the glucose-potassium ratio predict mortality in major burn patients? The glucose-to-potassium ratios of major burn patients at the time of initial hospitalization will be determined, and their relationship with mortality will be analyzed.

DETAILED DESCRIPTION:
Major burns, especially electrical burns, facial burns, inhalation burns, burns with large burn surface areas, and deep burns, have a high mortality risk. Early detection of this risk may be critical to reducing mortality rates. For this reason, trauma centers are working on rapid and effective prognostic markers. In trauma and stress situations, glucose levels rise while potassium levels fall due to increased catecholamines. The literature reports that hyperglycemia, also known as the glucose-potassium ratio, can rapidly and effectively predict morbidity and mortality in patients suffering from subarachnoid hemorrhage, pulmonary embolism, traumatic brain injury, or blunt abdominal trauma. Many publications show that increased glucose is associated with mortality and morbidity in critical illnesses and trauma. The isolated glucose-potassium ratio has a higher predictive ability for mortality and morbidity compared to glucose and potassium levels. In this study, investigators aimed to examine the prognostic value of the glucose-to-potassium ratio in participants with major burn trauma.

ELIGIBILITY:
Inclusion Criteria:

* All burns >40% of total body surface area (2nd degree or deeper)
* Burns with inhalation injury
* Burns >20% of total body surface area 3nd degree or deeper

Exclusion Criteria:

* First degree burns
* Patients have more than 24 hours since the onset of burn trauma
* Patients with diabetes mellitus
* Patients with chronic renal failure
* Patients taking potassium-modifying medication
* Patients with missing data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of patients of all age groups who were admitted to the burn center between May 2022 and May 2024 with 2nd degree and deeper burns of 40% and above total burn surface area, 3rd and 4th degree burns of 20% and above total burn surface area, and inhalation burns. Patients with missing data, patients with burn trauma of more than 24 hours since the onset of burn trauma, 1st degree burns, patients with diabetes mellitus or renal failure, and patients using potassium-regulating drugs were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Glucose-to-potassium ratio | 2 days
  The glucose-to-potassium ratio is calculated by dividing the participants' glucose values when they first apply to the hospital by their potassium values.

SECONDARY OUTCOMES:
Female/Male ratio | 2 days
  It is calculated by dividing the number of females by the number of males in the study population.
Mean percent of total body surface area burned | 2 days
  It is calculated by adding the total burn surface area percentage values of all patients and dividing by the number of participants.
Burn infection rate | 2 days
  The number of patients developing burn infection is calculated by dividing by the number of all participants.
Mortality rate | 2 days
  The mortality rate is calculated by dividing the number of patients who developed mortality by the number of all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Alpaslan Sahin, Assoc. Prof., Principal Investigator — Principal Investigator
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)